CLINICAL TRIAL: NCT02330107
Title: Effectiveness of Auriculotherapy on Lower Urinary Tract Symptoms in Elderly Men: A Randomized Controlled Feasibility Study.
Brief Title: Auriculotherapy on Lower Urinary Tract Symptoms in Elderly Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Lorna Suen, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-ZVD4
Record Dates: First submitted 2014-12-25; First posted 2015-01-01 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment arm 1 (Experimental): Subjects will receive MAT and placebo LA. The magnetic pellets will be applied to the six selected acupoints as detected by an acupoint finder. To achieve a blinding and placebo effect of the subject, the laser device will be switched to "power off" mode (i.e. deactivated laser) for acupoint "stimulation" before the application of MAT. Subjects will be asked to wear a pair of laser protective goggles to "blind" them during treatment.
  Interventions: Other: MAT & LAT
- Treatment arm 2 (Experimental): Subjects will receive a combined approach that includes the use of MAT and LA. A laser device (Pointer Pulse™) will be used in this study. This device has a wavelength of 650 nm, an average output power of 2.5 mW, an energy density of 1 minute with 0.54 J/cm2, and a pulse of 10 Hz, which is a common acceptable dosage for clinical use (King et al., 1990; Round et al., 2013). This application is a low-energy laser therapy (LLLT), in which the energy level emitted from the device is approximately comparable to a teaching pointer. A 1-minute treatment using the continuous mode of the device will be directly applied to the reactive region of each of the six selected acupoints on the ear. Laser protective goggles will be provided to the subjects and the researchers for eye protection.
  Interventions: Other: MAT & LAT
- Treatment arm 3 (Placebo Comparator): Subjects will serve as a placebo control and will receive LA at "power off" mode (i.e. deactivated laser) for acupoint "stimulation" before the application of plasters centred with a small portion of Junci Medulla (mimicking the MAT treatment).
  Interventions: Other: MAT & LAT

INTERVENTIONS:
Other: MAT & LAT — For MAT, the magnetic pellets will have ~200 gauss/pellet magnetic flux densities on average, with a diameter of 1.76 mm, to be put on the 6 selected acupoints of the ear.
  For LAT, a laser device (Pointer Pulse™) will be used in this study. This device has a wavelength of 650 nm, an average output power of 2.5 mW, an energy density of 1 minute with 0.54 J/cm2, and a pulse of 10 Hz. A 1-minute treatment using the continuous mode of the device will be directly applied to the reactive region of each of the six selected acupoints on the ear.

SUMMARY:
Lower urinary tract symptoms (LUTS) represent a widespread health problem that negatively affects the quality of life (QoL) of majority of the male aging population. Although LUTS are not life threatening, these symptoms include urinary retention, voiding difficulty, frequent feeling of urinary urgency, and nocturia, all of which negatively affect the daily functions, sleep quality, and sexual activities of patients. Despite the proven effectiveness of conventional pharmacological therapies, most men are reluctant to try these treatments because of perceived side effects and potential complications. Other non-invasive complementary treatments for LUTS should be explored because of the limitations of pharmacological therapy.

Auriculotherapy (AT), one of the approaches in traditional Chinese medicine, is a therapeutic method in which specific points in the auricle are stimulated to treat various physical disorders. AT is a specialized form of acupuncture in which the ear is viewed as a microsystem of the body. A minimally invasive measure of AT, instead of using needles, is adopted in this study to avoid pain induction.

This randomized controlled trial (RCT) aims to determine the effectiveness of AT in improving the conditions of the elderly with LUTS in terms of symptom relief, enhancing QoL, and improving sleep conditions. Male subjects, who are 60 years old or above and with moderate to severe LUTS, will be recruited.

Subjects in 'Treatment arm 1' will receive MAT and placebo LA on specific auricular points on one side of the ear during each treatment session. Subjects in 'Treatment arm 2' will receive LA and placebo MAT using low-energy laser applied to selected acupoints of the ear, and a plaster centred with a portion of Junci Medulla that mimics MAT treatment will also be given. Subjects in 'Treatment arm 3' will receive a combined approach (both MAT and LA). Subjects in the 'placebo arm' will serve as placebo controls. Six auricular acupoints that are considered to affect LUTS will be selected. Only one ear at a time will receive treatment. Thus, the ears will be treated alternately. The total treatment period will be four weeks. The experimental objects will be replaced every other day. Therefore, treatment will be performed thrice a week. Subjects will be assessed at baseline up to 3 months after the therapy. This study can advance our knowledge of complementary approaches to improve the LUTS conditions of the elderly population and the feasibility of AT among clients with LUTS in a future large-scale study.

DETAILED DESCRIPTION:
Research hypotheses:

1. Magneto-auriculotherapy (MAT) or laser auriculotherapy (LA) alone or use in combination are more effective than the control treatment in terms of symptom relief in male elderly patients suffering from LUTS.
2. MAT or LA alone or use in combination are more effective than the control treatment in terms of enhancement of QoL, and improvement of sleep conditions in male elderly patients suffering from LUTS.

Primary objective To investigate whether MAT or in combination with LAT are more effective than the control treatment in terms of symptom relief in male elderly patients suffering from LUTS.

Secondary objectives

1. To determine whether MAT or in combination with LAT are more effective than the control treatment in terms of enhancement of QoL, and improvement of sleep conditions in male elderly patients suffering from LUTS;
2. To assess the feasibility of using AT among LUTS patients in a future large-scale study, including the use of blinding, acceptance of treatment protocol, follow-up for repetitive testing, estimating effect size and attrition rate.
3. To compare the treatment effect and the feasibility of this study to be conducted in Hong Kong and China Mainland.

Research plan and methodology Design: This study is a randomized controlled and double-blinded feasibility trial.

Participants and settings.

In Hong Kong:

Subjects who are 60 years old or above will be recruited from the community centres or day care centres. The therapies will be administered either in the Integrative Health Clinic of the School of Nursing, The Hong Kong Polytechnic University, or in the elderly centres, depending on the subjects' convenience.

In China:

Subjects will be recruited by the Nursing College of Zhengzhou University. The inclusion and exclusion, therapy administration, and outcome measures will be identical with the study conducted in Hong Kong to facilitate comparison.

All therapies will be administered in a room assigned for research purposes. Only the researchers and the subject under treatment will be allowed to stay in the room during the therapy. A warning sign for laser radiation will be put up in a visible place outside the room for other workers or members of the elderly centres to see.

Groupings Group 1 (MAT & placebo LAT): Subjects will receive MAT. The magnetic pellets will have ~200 gauss/pellet magnetic flux densities on average, with a diameter of 1.76 mm (Figure 1). The experimental object will be applied to the six selected acupoints as detected by an acupoint finder. The Chinese Standard Ear-Acupoints Chart, which is recognized by the World Health Organization, is used to locate the reflective zones. These zones are as follows: angle of superior concha/prostate, kidney, bladder, ureter, external genitals, and internal genitals (Wang, Ceng, Wang, Lin & Wang, 1999). To achieve a blinding and placebo effect of the subject, the laser device will be switched to "power off" mode (i.e. deactivated laser) for acupoint "stimulation" before the application of MAT. Subjects will be asked to wear a pair of laser protective goggles to "blind" them during treatment.

Group 2 (Combined MAT & LAT): Subjects will receive a combined approach that includes the use of MAT and LA. A laser device (Pointer Pulse™) will be used in this study. This device has a wavelength of 650 nm, an average output power of 2.5 mW, an energy density of 1 minute with 0.54 J/cm2, and a pulse of 10 Hz, which is a common acceptable dosage for clinical use (King et al., 1990; Round et al., 2013). This application is a low-energy laser therapy (LLLT), in which the energy level emitted from the device is approximately comparable to a teaching pointer. A 1-minute treatment using the continuous mode of the device will be directly applied to the reactive region of each of the six selected acupoints on the ear. Laser protective goggles will be provided to the subjects and the researchers for eye protection (Figure 2).

Group 3 (Placebo MAT & placebo LAT): Subjects will serve as a placebo control and will receive LAT at "power off" mode (i.e. deactivated laser) for acupoint "stimulation" before the application of plasters centred with a small portion of Junci Medulla (mimicking the MAT treatment). Junci Medulla is the dried stem of the perennial plant that is soft in texture. It has been successfully adopted as a placebo in a previous study conducted by the PI because it does not induce any physical pressure on the acupoints of the ear (Suen et al., 2002a).

Experimental and control interventions Eligible subjects will be randomly and blindly allocated to one of the three groups, to be decided by a computer-generated randomised table. Restricted randomisation by blocking will be used to ensure approximately similar sample sizes for each group at any time during the trial according to equal proportion rule (1:1:1). The random allocation sequence will be managed by a specified research assistant (RA) who is not involved in this trial and is concealed to the assessors.

ELIGIBILITY:
The inclusion criteria are the following: (1) men aged 60 years old or above with LUTS for over two months and with an International Prostate Symptom Score (IPSS) of >=12 (moderate to severe LUTS symptoms) and (2) Maximum urinary flow rate (Qmax) of >=5 to <=15 ml/s with minimum voided urine >=125ml (Roberts, Lieber, Jacobson, Girman & Jacobsen, 2005; Roehrborn, 2005).

The exclusion criteria are the following: (1) patients who previously underwent or anticipated to receive minimal invasive therapies (e.g., transurethral microwave heat treatments and stent insertion) or surgical intervention of any kind (e.g., transurethral resection of the prostate, transurethral laser vaporization, and coagulation) within six months;(2) suffer from a psychiatric illness; (3) have prostate cancer history; (4) have chronic renal failure; (5) inability to understand instructions or give consent; and (6) suffering from aural injuries or infections.

For those who are receiving pharmacotherapy for BPH but can meet the inclusion criteria, they can be recruited into the study, but this has to be indicated in the data collection form.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
1. International Prostate Symptom Score (IPSS - Hong Kong Chinese Version 2) | collected at baseline up to 3 months after therapy
  This instrument will be used to collect information regarding the LUTS condition of the subjects. The instrument consists of seven Likert-scale questions [scores from 0 (not at all) to 5 (almost always)] that will address two aspects of LUTS. Three questions involve filling problems (daytime frequency and nocturnal urgency), and four questions assess voiding problems (emptying, intermittency, weak stream, and straining). The total IPSS score from the seven questions ranges from 0 to 35. The IPSS (Hong Kong Chinese version 2) has been recently validated and found to be a valid, reliable, and sensitive measure for assessing Chinese populations with LUTS (Cronbach's alpha coefficient = 0.71, ICC of the symptom questions = 0.80, ICC of the QoL = 0.70) (Choi et al., 2014). This tool will be set as the primary variable to indicate the actual effect size and continuously monitor the effectiveness of the treatments throughout the study.

SECONDARY OUTCOMES:
Maximum urinary flow rate (Qmax) | collected at baseline up to 3 months after therapy
  The participant will be asked to urinate into a special funnel connected to a portable uroflowmeter, which will measure the Qmax per second and help evaluate the severity of urinary obstruction.
2. Post-void residual urine test | collected at baseline up to 3 months after therapy
  The volume of urine (in mL) remaining in the bladder after voiding will be measured using a portable bladder scanner (BVI-9400) placed on the suprapubic region of the patient
Pittsburgh sleep quality index | collected at baseline up to 3 months after therapy
  This instrument will be used to collect data related to the sleep patterns of the subjects. The total PSQI score ranges from 0 to 21, and a PSQI score greater than 5 indicates poor sleep quality. The PSQI has been translated into 55 languages. Chong and Cheung (2012) validated the Cantonese PSQI and reported a high internal consistency of 0.75
Subjects' expectations towards therapy | collected at baseline up to 3 months after therapy
  A short questionnaire comprising six items is designed to assess patient's expectations towards the therapies that they will be receiving. Questions include which intervention that they think they have received, how strongly they believe that MAT or LA can help them manage their problem and how much faith they have in complementary therapies. The subjects will use a 10-point scale for most items. High scores would indicate high agreement or satisfaction with each item. The subjects will also be asked to describe their expectations for improvement of their LUTS without regarding to treatment using a 7-point Likert Scale with responses ranging from "completely gone" to "much worse". These items are adapted from existing literature (Kalauokalani et al., 2001; Molassiotis et al., 2013) and are modified for use in this study. This scale will be translated to Chinese and backward translation will be done in order to ensure the original meaning of the item is attained.
Patient satisfaction towards therapy | collected at baseline up to 3 months after therapy
  (1 item), for post-therapy evaluation only.
Other parameters | collected at baseline
  Socio-demographic characteristics include age, gender, body mass index, years of diagnosis (if known), TCM diagnosis differentiation, marital status, educational level, co-morbid illnesses, and current medications will be obtained. Other effects caused by therapy, such as allergic reactions to the skin due to the adhesive tape (for positioning the experimental objects), will also be evaluated after 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lorna KP Suen, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- The Neighbourhood Advice-Action Council, Hong Kong, Hong Kong